CLINICAL TRIAL: NCT06034548
Title: Diabetes and Hypertension Self Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1607202245
Record Dates: First submitted 2018-04-18; First posted 2023-09-13 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Intervention Model Description: RCT with wait-listed control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diabetes and hypertension self-management (Experimental): 12-week lifestyle and disease self-management
  Interventions: Behavioral: diabetes and hypertension self-management
- Control (No Intervention): Wait-list control

INTERVENTIONS:
Behavioral: diabetes and hypertension self-management — 12-weeks of 75 minutes of educational sessions
  Arms: diabetes and hypertension self-management

SUMMARY:
The purpose of this R15 project is to test the feasibility and effectiveness of a 12-week diabetes and hypertension self-management program using trained health coaches.

DETAILED DESCRIPTION:
West Virginia has high prevalence of comorbid diabetes and hypertension. Most diabetes self-management programs are hospital or clinic based and none are tailored to address the unique needs of rural WV adults with comorbid diabetes (T2DM) and hypertension (HTN). There is a critical need for new and creative community-based, culturally appropriate self-management programs in this medically underserved state. This study will use a wait-listed randomized control trial (RCT) design, using evidence-based interventions, to improve patient self-management behaviors and health outcomes (HbA1c and BP). Eligible adults with comorbid T2DM and HTN will be randomized with a 1:1 ratio to the immediate diabetes and hypertension self-management program (DHSMP; n=35) or to 6-month wait-listed control group (N=35), based on an allocation sequence generated by the biostatistician using a randomly varying block randomization method to ensure equal distribution among treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults >= 18 years of age;
* co-occurring diagnosis of T2DM and HTN;
* body mass index >= 25.0
* willing to be randomized and complete all assessments.

Exclusion Criteria:

* currently pregnant or breastfeeding;
* diagnosed with a severe mental illness;
* have any condition that requires physical activity limitations or is contraindicated for the Dietary Assessment to Stop Hypertension (DASH) diet;
* inability to complete the study protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes - A1c | 6 months after enrollment
  The difference in A1c between baseline and end of program.
Clinical outcomes - BP | 6 months after enrollment
  The difference in BP (systolic and diastolic) between baseline and end of program.

SECONDARY OUTCOMES:
Behavioral outcome - healthy eating plan; questions | 6 months after enrollment
  Dietary analysis will be based on following a healthy eating plan at baseline and completion of the Program. All participants will be assessed regarding the number of days they followed a healthful eating plan using a survey question from the Summary of Diabetes Self-care activities measure by Toolbert et al., Diabetes Care, 2000. "How many of the last SEVEN DAYS have you followed a healthful eating plan?" 0 1 2 3 4 5 6 7. Changes in mean number of days followed a healthy eating plan will be assessed at baseline and at the completion of the program.
Behavioral outcome - exercise; questions | 6 months after enrollment
  All participants will be assessed regarding the number of days they exercise using two survey questions from the Summary of Diabetes Self-care activities measure by Toolbert et al., Diabetes Care, 2000. The description of the questions are as follow: Q1. "On how many of the last SEVEN DAYS did you participate in at least 30 minutes of physical activity? (please list the total minutes of continuous activity, including walking)" 0 1 2 3 4 5 6 7 & Q2. "On how many of the last SEVEN DAYS did you participate in a specific exercise session (such as swimming, walking, biking) other than what you do around the house or as part of your work?" 0 1 2 3 4 5 6 7). The total exercise score will be calculated by the mean number of days for the two questions). Changes in mean number of days exercised will be assessed at baseline and at the completion of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjita Misra, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No